CLINICAL TRIAL: NCT02500329
Title: Effect of Gemigliptin or Acarbose on Endothelial Function in Type 2 DM Patients (GetUp Trial)
Brief Title: Effect of Gemigliptin or Acarbose on Endothelial Function in Type 2 DM Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Min Kyong Moon, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRMH 26-2014-124
Record Dates: First submitted 2015-07-12; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Endothelial Function; Type 2 Diabetes; Gemigliptin; Acarbose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; Acarbose

ARMS (2):
- gemigliptin (Experimental): gemigliptin for 4 weeks
  Interventions: Drug: Gemigliptin
- acarbose (Active Comparator): acarbose for 4 weeks
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Gemigliptin — Gemigliptin for 4 weeks
  Arms: gemigliptin
Drug: Acarbose — Acarbose for 4 weeks
  Arms: acarbose

SUMMARY:
This is a phase 4, single center, randomized, open-labeled study. The primary objective of the study is to compare effect of gemigliptin and acarbose on endothelial function.

Subjects are randomized to gemigliptin or acarbose group and maintained intial treatment for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age: 20-80yrs
* patients with type 2 diabetes (duration of diabetes >=3 months)
* HbA1c :>7.0 and <=9.0% on metformin monotherapy
* no changes on medications during recent 3 months.

Exclusion Criteria:

* patients with type 1 diabetes
* history of medications including α-glucosidase inhibitor, glinide, GLP-1 analogue, other DPP-4 Inhibitors, or insulin during recent 3 months.
* history of acute diabetic complication, acute coronary events, or coronary bypass surgery/interventions during recent 6 months.
* patients with congestive heart failure (NYHA II~IV) or clinically significant ventricular arrhythmia
* serum ALT or AST> 2.5 x upper normal range
* serum direct bilirubin > 1.3 x upper normal range
* serum creatinine > (men) 1.5 mg/dL, (women)>1.4 mg/dL
* smoker
* pregnant women, or breast-feeding women
* medication with acetylsalicylic acid or vitamin K antagonist

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
endothelial function (reactive hyperemic index) | 4 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose | 4 weeks
Postprandial 2hour glucose | 4 weeks
Glycated albumin | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Min Kyong Moon, Principal Investigator — Boramae medical center, 20 Boramae-ro 5-gil,Dongjak-Gu,Seoul 156-707, Korea
Locations (1):
- Boramae medical center, Seoul, South Korea